CLINICAL TRIAL: NCT00578825
Title: A Multi-centre, Double-blinded, Randomized, Placebo-controlled Trial on the Efficacy and Safety of Lopinavir / Ritonavir Plus Ribavirin in the Treatment of Severe Acute Respiratory Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KW/FR/04-009; HARECCTR0500028; NTWC/CREC/349/05
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: Severe acute respiratory syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Lopinavir; Ritonavir; Ribavirin

INTERVENTIONS:
Drug: Lopinavir / Ritonavir plus Ribavirin

SUMMARY:
The study aims to examine whether the combination of Lopinavir/Ritonavir plus Ribavirin for treatment of severe acute respiratory syndrome (SARS) is superior to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18 with a diagnosis of SARS and with valid consent will be recruited.

Exclusion Criteria:

* Subjects with medical conditions that makes the prescription of study medications unsafe are excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)

PRIMARY OUTCOMES:
Development of severe SARS | Any time during the acute illness

SECONDARY OUTCOMES:
Adverse events | Throughout the illness period
SARS-CoV Viral load | Throughout the illness period
Immunological profile | Throughout the illness period

CONTACTS AND LOCATIONS:
Overall Officials: Wai Cho Yu, Dr, Principal Investigator — Department of Medicine & Geriatrics, Princess Margaret Hospital
Locations (9):
- China (9):
  - Department of Health, Hong Kong
  - Kowloon Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong, Hong Kong
  - The University of Hong Kong, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - United Christian Hospital, Hong Kong